CLINICAL TRIAL: NCT02388958
Title: Weight Changes During and After Pregnancy in Women With Gestational Diabetes
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Rosette Chakkalakal, Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 140295; P30DK092986 (NIH)
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Gestational Diabetes Mellitus
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women with GDM
- Women without GDM

SUMMARY:
Gestational diabetes mellitus (GDM) is associated with short-term and long-term complications for infants and mothers. The management of GDM during pregnancy focuses on reducing risks to the infant associated with hyperglycemia. The postpartum management of GDM focuses on reducing maternal risk of developing type 2 diabetes (T2DM). A diagnosis of GDM identifies up to 31% of parous women who will eventually develop T2DM and approximately 50% of women diagnosed with GDM will develop T2DM in the first 5 years postpartum. The perceived risk of developing short-term and/or long-term complications of GDM may influence women's likelihood of engaging in diet modification, the mainstay of treatment of GDM, both during and after pregnancy. If sustained after delivery, diet modifications introduced as treatment for GDM could affect maternal weight changes during and after pregnancy, which could in turn affect T2DM risk. It is unknown if and how women with GDM differ in their perceived risk of developing T2DM, dietary choices, or weight gain (and retention) during versus after pregnancy. Therefore, the project proposed in this application seeks to (1) characterize the perceived risk of developing T2DM among women with GDM during and after pregnancy, (2) characterize dietary choices of women with GDM during and after pregnancy, and (3) characterize weight changes of women with GDM during and after pregnancy as compared to women without GDM.

ELIGIBILITY:
Inclusion Criteria for women with GDM:

* Patient is currently pregnant with a singleton pregnancy.
* Laboratory confirmed diagnosis of GDM between weeks 24-28 gestation.
* Patient is receiving routine prenatal care at Vanderbilt University Medical Center.

Inclusion Criteria for women without GDM:

* Patient is currently pregnant with a singleton pregnancy.
* Patient does not have GDM based on non-fasting and/or fasting GTT results.
* Patient is receiving routine prenatal care at Vanderbilt University Medical Center.

Exclusion Criteria for both cohorts:

* Diagnosis of type 1 or type 2 diabetes prior to pregnancy.
* Diagnosis of GDM prior to 20 weeks gestation.
* Patient does not speak English.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All women receiving prenatal care at Vanderbilt University Medical Center who do not already carry a diagnosis of type 1 or type 2 diabetes are screened for GDM between weeks 24-28 of pregnancy with a non-fasting 50-gram glucose tolerance test (GTT). Blood glucose values greater than or equal to 140 on this screening test are considered positive. Women with a positive screening test undergo a diagnostic fasting 100-gram 3-hour GTT. GDM is diagnosed if a woman has 2 or more abnormal values on the 3-hour GTT (abnormal values are fasting blood glucose greater than or equal to 95, 1-hour blood glucose greater than or equal to 180, 2-hour blood glucose greater than or equal to 155 and/or 3-hour blood glucose greater than or equal to 140). By reviewing the electronic medical record of women with singleton pregnancies undergoing GTT on a weekly basis, we will identify women with and without GDM.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Postpartum weight change measured in kilograms | 6 months (change in weight from the time of delivery to 6 months postpartum)

SECONDARY OUTCOMES:
Rate of pregnancy weight gain prior to GDM diagnosis measured in kilograms per week | 24-28 weeks
Rate of pregnancy weight gain after GDM diagnosis measured in kilograms per week | 10-16 weeks
Change in perceived risk of developing diabetes during versus after pregnancy measured with the Risk Perception Survey for Developing Diabetes (RPS-DD) | 10 months
Change in dietary choices during versus after pregnancy measured with the Personal Diabetes Questionnaire | 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosette Chakkalakal, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States